CLINICAL TRIAL: NCT01335633
Title: Psychometric Validation of Cognitive Endpoints
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, John DeLuca, Vice President of Research, Kessler Foundation
Other Study IDs: 691-11 PVCE
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Sclerosis
Keywords: MS; Neuropsychological tests
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will entail cognitive assessment of a single cohort of patients with Multiple Sclerosis. Each subject will be assessed twice, approximately 45 days apart. There will be no intervention or control group. Each participant will have a caregiver capable of responding to a brief report of observations regarding neuropsychological skills and abilities in the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old (inclusive).
* History of Relapsing-Remitting or Secondary Progressive Multiple Sclerosis
* Physically able to see the testing materials and complete the tests
* Have a family member or caregiver who is capable of consent and willing to complete the MSNQ-Informant questionnaire.

Exclusion Criteria:

* A history of treated or untreated severe mental illness or diagnosis of major depression prior to MS onset.
* Untreated major depression or untreated anxiety disorder.
* History of Attention Deficit/Hyperactivity Disorder, Developmental Learning - Disorder including Mental Retardation.
* History of traumatic brain injury with intracranial bleed, stroke, Alzheimer's disease, Parkinson's disease, Motor Coordination Disorder or other neurologic illness. I understand that if the Investigator believes this would interfere with successful completion of the protocol, I will be excluded.
* A clinically significant relapse within the past 2 months. I have had a serious infection (e.g., pneumonia, septicemia) within the 2 month.
* History of drug or alcohol abuse (as defined by the Investigator) within 1 year prior to Study Day 1.
* Active bacterial or viral infection.
* Use of marijuana within 2 months prior to Study Day 1or at any time during the study
* Alcohol consumption within 24 hours of either test session.
* Unable to comply with study requirements.
* Expected survival time of less than 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, Ph.D., Principal Investigator — Kessler Foundation
Locations (4):
- United States (4):
  - Holy Name Hospital Multiple Sclerosis Center, Teaneck, New Jersey
  - Kessler Foundation, West Orange, New Jersey
  - University at Buffalo, Buffalo, New York
  - Lauren S. Caruso, White Plains, New York